CLINICAL TRIAL: NCT04347096
Title: Effects and Cost-effectiveness of an mHealth Intervention to Improve Diet, Physical Activity and Sedentary Behavior Among Sedentary Workers
Brief Title: Effects of an mHealth Intervention to Improve Health Behaviors Among Sedentary Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); China Medical University, Taiwan (Other)
Responsible Party: Principal Investigator, Lin, Yun-Ping, Associate Professor, China Medical University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CRREC-109-017
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2020-07

CONDITIONS: Intervention Study; Health Behavior
Keywords: Sedentary workers; Healthy diet; Physical activity; Mobile Health; Web app; Cardiometabolic risk biomarkers; Work productivity; Cost-effectiveness
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mHealth Intervention (Experimental): The mHealth intervention group will have access to the Internet for using a newly developed Simple health web app and receive an activity tracker. The web app users are required to: (1) wear an activity tracker every day; (2) set goals of daily stand-up, physical activity, and healthy eating bi-weekly; (3) record stand-up, physical activity, and healthy eating behaviors daily; (4) set reminders to stand-up and record health behaviors; and (5) read educational and motivational tools. After completing the behavioral record, the personal advice will automatically provide to encourage, motivate and support the user. Moreover, the user will be able to look at his/her personal and team health ranking.
  Interventions: Behavioral: mHealth Intervention
- Control Intervention (Other): The control intervention group will only receive educational tools (usual care).
  Interventions: Behavioral: Control Intervention

INTERVENTIONS:
Behavioral: mHealth Intervention — The mHealth Intervention will provide sedentary workers with evidence-based information on diet, physical activity and sedentary behavior, and tailored feedback on their responses to daily records. Key features of this intervention will include individualized feedback and multimedia presentation in the form of web app. The intervention group will also receive a reliable device for wireless physical activity tracking for monitoring step counts.
  The web app will consist of seven major components: (1) daily healthy eating goals and records; (2) daily physical activity goals and records; (3) daily stand-up goals and records; (4) advice and reminder; (5) educational and motivational tools; (6) personal and team health ranking; and (7) online social network. In addition, the intervention will be enhanced with follow-up booster coaching calls bi-monthly at 2, 4, 6, 8 months after the 12-week intervention.
  Arms: mHealth Intervention
Behavioral: Control Intervention — The control intervention group will receive educational tools, which will provide knowledge on benefits of physical activity and healthy eating, health risks of sitting and unhealthy diets, and recommendations on physical activity and a balanced healthy diet for good health.
  Arms: Control Intervention

SUMMARY:
Background: Studies have shown the negative impact of physical inactivity, sedentary and unhealthy eating behavior on worker health and productivity. Sedentary workers are at greater risk of developing chronic diseases due to these behavioral risk factors. The literature moderately supports mHealth interventions for promoting physical activity and healthy diets. However, there is a dearth of research on mHealth interventions targeting the clustering of physical activity, sedentary and dietary behavior among sedentary workers in the occupational setting. Furthermore, there is a lack of evidence on its long-term sustainability and cost-effectiveness on health behaviors as well as health-related and work- related outcomes.

Purpose: To evaluate a 12-week theory-driven, tailored mHealth intervention for improving diet, physical activity and sedentary behavior among sedentary workers. Three specific aims are to: (1) determine intervention participants' perceptions of and engagement with the mHealth program components to understand intervention effects by surveys and focus groups; (2) determine the effectiveness of the mHealth intervention compared to usual care; and (3) determine the cost-effectiveness of the mHealth intervention compared to usual care, using incremental cost-effectiveness ratios (ICERs).

Methods: This is a three-year research project. Year 1 is mHealth intervention delivery and evaluation using a quasi-experimental design. Concepts of social cognitive theory of self-regulation and self-efficacy and an ecological model provide the theoretical foundation for the intervention. Year 2 will be primarily to evaluate the intervention. Year 3 will be primarily an international comparison of cost-effectiveness of mHealth interventions to improve diet, physical activity and sedentary behavior for employees.

A total of 100 sedentary workers (50 per condition) will be recruited from two workplaces. The intervention group will have access to the Internet for using a newly developed Simple health web app and receive an activity tracker. A sample of 100 is required to detect differences in primary outcomes: cardiometabolic risk biomarkers, productivity loss, body composition, physical activity, sedentary behavior, and dietary behavior; and secondary outcomes: self-report self-efficacy and self-regulation, at baseline, 3-, 12-, and 24-month follow up. Generalized estimating equations (GEE) will be used to examine intervention effects over time.

DETAILED DESCRIPTION:
The Simple health web app will consist of six major components: (1) daily healthy eating goals and records; (2) daily physical activity goals and records; (3) daily stand-up goals and records; (4) advice and reminder; (5) educational and motivational tools; and (6) personal and team health ranking.

ELIGIBILITY:
Inclusion Criteria:

1. Full-time employees with sedentary occupations that involve sitting most of the time.
2. Age 20 years and older.
3. No physical limitations that would prevent them from performing physical activity.
4. Has access to the Internet.

Exclusion Criteria:

1. Part-time employees.
2. Has an expected absence from work for more than two weeks or an expected relocation to another workplace within the next 3 months.
3. Pregnant or planning to get pregnant within the next 3 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Objectively measured physical activity | Changes from baseline objectively measured physical activity at 3-, 12-, and 24-month
  Physical activity will be objectively measured by the wrist-worn Fitbit Charge 3 (3-axis accelerometer)
Self-report physical activity | Changes from baseline self-report physical activity at 3-, 12-, and 24-month
  Physical activity will be assessed by International Physical Activity Questionnaire (IPAQ)-Taiwan short form
Objectively measured dietary behavior | Changes from baseline objectively measured dietary behavior at 3-, 12-, and 24-month
  Dietary behavior will be objectively measured with 3-day food photography
Self-report dietary behavior | Changes from baseline self-report dietary behavior at 3-, 12-, and 24-month
  Dietary behavior will be assessed by the Healthy Eating Behavior Inventory (HEBI)
Occupational sitting and physical activity | Changes from baseline occupational sitting and physical activity at 3-, 12-, and 24-month
  Occupational sitting and physical activity will be assessed by the Occupational Sitting and Physical Activity Questionnaire (OSPAQ)
Work productivity | Changes from baseline work productivity at 3-, 12-, and 24-month
  Work productivity will be measured by Work Limitation Questionnaire (Taiwan) short-form (WLQ-SF)
Fasting blood glucose | Changes from baseline fasting blood glucose at 3-, 12-, and 24-month
  Fasting blood glucose will be measured by collecting fasting blood samples in the morning
Fasting insulin | Changes from baseline fasting insulin at 3-, 12-, and 24-month
  Fasting insulin will be measured by collecting fasting blood samples in the morning
Total cholesterol | Changes from baseline total cholesterol at 3-, 12-, and 24-month
  Total cholesterol will be measured by collecting fasting blood sample in the morning
Low-density lipoprotein (LDL) cholesterol | Changes from baseline LDL cholesterol at 3-, 12-, and 24-month
  LDL cholesterol will be measured by collecting fasting blood sample in the morning
High-density lipoprotein (HDL) cholesterol | Changes from baseline HDL cholesterol at 3-, 12-, and 24-month
  HDL cholesterol will be measured by collecting fasting blood sample in the morning
Triglycerides | Changes from baseline triglycerides at 3-, 12-, and 24-month
  Triglycerides will be measured by collecting fasting blood samples in the morning
Blood pressure | Changes from baseline blood pressure at 3-, 12-, and 24-month
  Blood pressure will be measured twice per person via an automated sphygmomanometer using the right arm and an appropriately sized cuff. A third measurement will be taken if the systolic BP differs by >10 mmHg or the diastolic BP by >6 mmHg.
Weight | Changes from baseline weight at 3-, 12-, and 24-month
  Weight will be measured by ioi 353 body composition analyzer (JAWON MEDICAL)
Abdominal circumference | Changes from baseline abdominal circumference at 3-, 12-, and 24-month
  Abdominal circumference will be measured by ioi 353 body composition analyzer (JAWON MEDICAL)
Percent body fat | Changes from baseline percent body fat at 3-, 12-, and 24-month
  Percent body fat will be measured by ioi 353 body composition analyzer (JAWON MEDICAL)
Soft lean mass | Changes from baseline soft lean mass at 3-, 12-, and 24-month
  Soft lean mass will be measured by ioi 353 body composition analyzer (JAWON MEDICAL)
Visceral fat area | Changes from baseline visceral fat area at 3-, 12-, and 24-month
  Visceral fat area will be measured by ioi 353 body composition analyzer (JAWON MEDICAL)

SECONDARY OUTCOMES:
Self-efficacy for reducing sitting | Changes from baseline self-efficacy for reducing sitting at 3-, 12-, and 24-month
  Self-efficacy for reducing sitting will be assessed by the self-efficacy for reducing sitting scale
Self-efficacy for physical activity | Changes from baseline self-efficacy for physical activity at 3-, 12-, and 24-month
  Self-efficacy for physical activity will be assessed by the self-efficacy for physical activity scale
Self-efficacy for healthy eating | Changes from baseline self-efficacy for healthy eating at 3-, 12-, and 24-month
  Self-efficacy for healthy eating will be assessed by the self-efficacy for healthy eating scale
Self-regulation of sitting less and moving more | Changes from baseline self-regulation of sitting less and moving more at 3-, 12-, and 24-month
  Self-regulation of sitting less and moving more will be assessed by the self-regulation for sitting less and moving more scale
Self-regulation of eating behaviour | Changes from baseline self-regulation of eating behaviour at 3-, 12-, and 24-month
  Self-regulation of eating behaviour will be assessed by the Self-Regulation of Eating Behaviour Questionnaire

OTHER OUTCOMES:
Cost-effectiveness | At 3-, 12-, and 24-month
  Cost-effectiveness will be assessed by constructing the incremental cost-effectiveness ratio (ICER)

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Ping Lin, PhD, Principal Investigator — China Medical University, Taiwan
Locations (1):
- China Medical University, Taichung, N/A = Not Applicable, Taiwan

REFERENCES:
- [Derived] Lin YP, Lu SH, Lee KC, Ma WF, Ho YF, Liao WC, Yang HT, Hong O. Short-Term Effects of a Mobile Health Intervention on Healthy Behaviors and Cardiometabolic Health in Sedentary Employees: A Quasi-Experimental Study. JMIR Mhealth Uhealth. 2026 Jan 22. doi: 10.2196/70074. Online ahead of print. PMID 41620395